CLINICAL TRIAL: NCT02091947
Title: Efficacy of Functional Magnetic Stimulation in Urinary Incontinence
Acronym: FMS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: vghtpe user (Other Government)
Responsible Party: Sponsor-Investigator, vghtpe user, Po-Yi Tsai MD, Taipei Veterans General Hospital, Taiwan
Organization: Taipei Veterans General Hospital, Taiwan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201010015OB
Record Dates: First submitted 2014-03-11; First posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Incontinence
Keywords: FMS; Urine incontinence
MeSH Terms: conditions — Nocturnal Enuresis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): Real FMS, 5 Hz, 20 minutes per day, for 10 weekdays.
  Interventions: Device: FMS (Magstim rapid2)
- sham group (Sham Comparator): sham FMS, 5 Hz, 20 min per day, for 10 weekdays.
  Interventions: Device: FMS (Magstim rapid2)

INTERVENTIONS:
Device: FMS (Magstim rapid2) — 5 Hz FMS, over bilateral sacral roots.

SUMMARY:
Functional Magnetic Stimulation (FMS) appears to modulate autonomic and somatic nervous systems that innervate the lower urinary tract. Stimulation of the pudendal afferent nerve near the third sacral root induces relaxation of the detrusor muscles and reinforcement of urethral sphincter. Some preliminary studies had indicated the positive effect of FMS on stress urinary incontinence. Investigators aimed to evaluate the immediate and long-term effect of this method on stress urinary incontinent patients.

DETAILED DESCRIPTION:
5 Hz repetitive magnetic stimulation was applied over bilateral sacral roots for 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Urine incontinence refractory to traditional treatment

Exclusion Criteria:

* Arrhythmia, pacemaker implantation

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-11; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Symptom scoring on Urge-Urinary Distress Inventory questionnaire | up to 5 months

SECONDARY OUTCOMES:
Cystometry and stress urethral pressure profile as measures of objective incontinence improvement | up to 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yi Tsai, MD, Principal Investigator — Dep of PMR, Taipei VGH
Locations (1):
- Taipei Veteran General Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Tsai PY, Wang CP, Hsieh CY, Tsai YA, Yeh SC, Chuang TY. Long-term sacral magnetic stimulation for refractory stress urinary incontinence. Arch Phys Med Rehabil. 2014 Dec;95(12):2231-8. doi: 10.1016/j.apmr.2014.07.010. Epub 2014 Jul 27. PMID 25073008